CLINICAL TRIAL: NCT06380816
Title: A Cancer Research UK Phase I/II Trial to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of UCB4594 Alone and in Combination With Anti-cancer Treatments in Participants With Advanced Malignancies
Brief Title: A Phase I/II Trial of UCB4594 in Participants With Advanced Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/24/001; ISRCTN26628699 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2024-03-27; First posted 2024-04-24 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumours; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Renal Cell (Clear Cell Only); Esophageal Neoplasms; Stomach Neoplasms (Excluding Gastrointestinal Stromal Tumors); Uterine Cervical Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms
Keywords: HLA-G; Monoclonal Antibody; Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Carcinoma; Esophageal Neoplasms; Stomach Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Module A (UCB4594 monotherapy dose escalation) (Experimental): Participants with advanced solid tumours from tumour types with known high levels of HLA-G expression (as reported in the literature) will be recruited.
  Interventions: Drug: UCB4594
- Module B (UCB4594 monotherapy expansion) (Experimental): Participants with a specific tumour type where HLA-G expression is more prevalent may be recruited to receive UCB4594 monotherapy.
  Interventions: Drug: UCB4594

INTERVENTIONS:
Drug: UCB4594 — Participants will receive UCB4594 as an intravenous infusion once every 3 weeks for up to 18 cycles, with each cycle lasting 21 days (~1 year).

SUMMARY:
This clinical trial is looking at UCB4594. This is the first time the drug is being tested in humans. UCB4594 is a type of drug called a monoclonal antibody. It has been designed to work by targeting a protein called human leucocyte antigen G (HLA-G) that is found in high levels on some cancer cells. By attaching itself to this protein it may help the immune system to attack and kill the cancer cells.

The four main aims of the clinical trial are to find out:

1. The best dose of UCB4594 that can be given safely to participants in the trial.
2. What the side effects of UCB4594 are and how they can be managed.
3. What happens to UCB4594 inside the body and how it affects cancer cells.
4. Whether UCB4594 can cause cancer to shrink.

DETAILED DESCRIPTION:
What does the study involve?

This clinical trial is split into two phases.

Phase I (Module A) is the 'dose escalation' phase. This is where small groups of participants receive UCB4594 at a certain dose level starting with a low dose level. After reviewing the results obtained at each dose level, it will be decided whether or how much to increase the dose for the next group of participants. This part of the study aims to find the best dose to give that does not cause too many side effects.

Phase II is the 'dose expansion' phase. This starts when the dose escalation phase has worked out the best dose of UCB4594 to give. In this part of the trial UCB4594 will be given alone (Module B) or in combination with other anti-cancer drugs (Module C). This will allow us to find out more about how the drug is working and whether UCB4594 affects cancer. Details for Module C of the dose expansion phase will be added when the types of cancer and anti-cancer drugs are defined.

What are the possible benefits and risks of participating?

UCB4594 is a new drug that has never been given to humans before. Possible risks and benefits are based on laboratory tests and experience with similar drugs but there is not yet any information about the effects of UCB4594 in humans. Participants in the trial will be monitored closely to find out the effects of UCB4594.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed and dated) informed consent and capable of co-operating with investigational medicinal product (IMP) administration and follow-up
2. Participant population: Histologically or cytologically proven advanced solid tumours (as specified below), refractory to conventional treatment, or for which no conventional therapy is considered appropriate by the Investigator or is declined by the participant. Module A (dose escalation): Tumour types which have shown high levels of human HLA-G expression (as reported in the literature): head and neck squamous cell carcinoma, non-small cell lung cancer, colorectal cancer, triple-negative breast cancer, renal cell cancer (clear cell only), oesophago-gastric cancer (excluding gastrointestinal stromal tumour), cervical cancer, ovarian cancer, pancreatic cancer. N.B. Participants with small cell type cancers on histology/cytology are excluded. Pre-treatment biopsies are mandatory for all participants. Paired biopsies will be mandatory for participants from doses of 30 mg and higher. Participants must have disease amenable to biopsy (excluding bone metastases) as deemed safe by the Investigator
3. Measurable disease, according to RECIST v1.1
4. Life expectancy of at least 12 weeks
5. Eastern Cooperative Oncology Group performance status of 0 or 1
6. Haematological and biochemical indices within defined ranges. These measurements should be performed to confirm the patient's eligibility to participate in the trial
7. Aged 18 years or over at the time consent is given. Participants aged 16-17 years may be eligible for recruitment to the backfill cohorts in dose escalation once adequate safety and toxicity data have been established in participants aged 18 years or over. All relevant data will be reviewed and a decision on the inclusion of participants aged 16-17 years will be made by the Trial Management Group

Exclusion Criteria:

1. Radiotherapy (except palliative), endocrine therapy (unless for non-malignant disease), chemotherapy, targeted therapy or immunotherapy, or any other IMPs during the previous 4 weeks or 5 half-lives (whichever is shorter) before the first dose of IMP
2. Ongoing toxicity of previous treatments >CTCAE Grade 1 (except alopecia of any grade, stable Grade 2 peripheral neuropathy or hormone-replacement therapy (HRT)-managed endocrine disorders)
3. Patients with rapidly progressing / symptomatically deteriorating brain/leptomeningeal metastases/untreated brain metastases are excluded. Patients with previously treated brain metastases are eligible if they haven't had a seizure or a clinically significant change in neurological status or required steroids in the last 2 weeks
4. Pregnant or breastfeeding female patients (or planning to breastfeed)
5. Women of childbearing potential. However, those not already pregnant or breastfeeding (or who discontinue breastfeeding) and meet the following are eligible:

   5.1. Have a negative serum pregnancy test within 7 days before enrolment and either:

   5.2.1. Agree to a form of highly effective contraception plus a barrier method, or

   5.2.2. Agree to sexual abstinence

   Effective from the negative pregnancy test, throughout the trial and for 10 months after the last dose of UCB4594
6. Male patients with partners of childbearing potential. However, patients who meet the following are eligible:

   6.1. Agree to a barrier method of contraception or sexual abstinence

   6.2. Males with pregnant or breastfeeding partners must use barrier method contraception to prevent exposure of the foetus or neonate

   6.3. Non-vasectomised males must also ensure any partner of childbearing potential uses highly effective contraception or agrees to sexual abstinence

   Effective from the date of the first dose of UCB4594, throughout the trial and for 5 months after the last dose of UCB4594 N.B. Males must refrain from donating sperm for the same period
7. Surgery from which the patient has not yet recovered
8. High medical risk because of non-malignant systemic disease, including serious or uncontrolled infection (requiring intravenous antibiotics) or unexplained fever >38°C within 2 weeks prior to the first dose of UCB4594
9. Known to be serologically positive for hepatitis B virus, hepatitis C virus or human immunodeficiency virus
10. Active or suspected autoimmune disease, or any history of autoimmune condition that required systemic corticosteroids or immunosuppressive agents. Patients who have ever had a transplant are excluded. This does not apply to patients with: vitiligo, alopecia, or type I diabetes mellitus, psoriasis not requiring chronic systemic immunosuppressive treatment within the past 2 years, stable autoimmune-mediated hypothyroidism on HRT, and Raynaud's syndrome
11. Are being treated with escalating or supraphysiologic doses of corticosteroids or immunosuppressive agents. Participants with immunotherapy-related hypophysitis adequately treated with physiologic doses of steroids are not excluded. Use of topical, ophthalmic, inhaled, intermittent steroid injections, and intranasal corticosteroids are permitted
12. Hypersensitivity to the ingredients/excipients (including polysorbate 80) in UCB4594
13. History of significant toxicities from treatment of immune checkpoint inhibitors (CPIs) that necessitated permanent discontinuation (Patients who started on combination CPI [e.g., ipilimumab/nivolumab] and had toxicity requiring discontinuation of one CPI [e.g., continued with nivolumab single agent] are not excluded)
14. History of Grade ≥3 infusion-related reaction to monoclonal antibodies or similar drugs
15. Prior treatment with HLA-G, immunoglobulin-like transcript (ILT)2 or ILT4-targeting drug
16. Live, attenuated vaccine within 28 days prior to the first dose of IMP
17. Increased risk due to tumour flare (e.g., an initial increase in tumour size that may lead to obstruction of airways, etc)
18. Significant active pulmonary disease or condition at screening, including:

    18.1. Lymphangitis carcinomatosa

    18.2. History of interstitial lung disease or pulmonary fibrosis

    18.3. History of pulmonary inflammatory disease
19. Evidence of bleeding diathesis
20. Significant cardiovascular disease, defined as a history of: congestive heart failure requiring therapy or left ventricular ejection fraction <40%, unstable angina pectoris or myocardial infarction within 6 months prior to entry, or current poorly controlled angina (symptoms weekly or more), clinically significant cardiac arrhythmia within 6 months prior to entry (asymptomatic atrial fibrillation or asymptomatic first-degree heart block permitted), or myocarditis. Presence of symptomatic or severe valvular heart disease. Baseline QT interval corrected by Fridericia >450 msec for males and >470 msec for females on triplicate electrocardiogram is ineligible
21. Participant in or plans to join another interventional trial
22. Other current malignancies. Cancer survivors who have undergone potentially curative therapy for prior malignancy with no evidence of disease for 3+ years are eligible
23. Any other condition that, in the Investigator's opinion, means the trial is not in the patient's best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 dose (RP2D) of UCB4594 | From Day 1 (date of first dose of UCB4594) up to Day 21.
  The RP2D will be the dose(s) of UCB4594 (in units of mg) selected for further evaluation and will be determined based on the maximum tolerated dose or maximum administered dose (MTD/MAD) and all available safety, efficacy, pharmacokinetic (PK) and pharmacodynamic data (all modules - dose escalation [module A], monotherapy dose expansion [module B] and any combination modules [module C]).
Frequency of adverse events (AEs) considered at least possibly related to UCB4594 (up to 18 cycles). | From time of informed consent up to 12 months
  AE data will be collected for UCB4594 (all modules) and/or other anti-cancer treatments (Module C), and the number of Grade 3, 4 and 5 AEs at least possibly related to UCB4594 (all modules) and/or other anti-cancer treatments (Module C) for up to 18 cycles (~12 months) of dosing determined. AEs, including relatedness, seriousness and severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, will be assessed by the Investigator.

SECONDARY OUTCOMES:
Number of patients achieving a complete response (CR)/immune CR (iCR) or partial response (PR)/immune PR (iPR) to UCB4594 (all modules). | From baseline radiological disease assessment up to 13 months.
  Number of patients achieving a CR/iCR or PR/iPR to UCB4594 (all modules) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 and immune RECIST (iRECIST).
Maximum concentration of UCB4594 (monotherapy modules; Modules A and B). | From Day 1 (date of first dose of UCB4594) up to 13 months.
  UCB4594 concentrations will be measured in serum.
Minimum concentration of UCB4594 (monotherapy modules; Modules A and B). | From Day 1 (date of first dose of UCB4594) up to 13 months.
  UCB4594 concentrations will be measured in serum.
Area under the curve of UCB4594 (monotherapy modules; Modules A and B). | From Day 1 (date of first dose of UCB4594) up to 13 months.
  UCB4594 concentrations will be measured in serum.
Steady state volume of distribution of UCB4594 (monotherapy modules; Modules A and B). | From Day 1 (date of first dose of UCB4594) up to 13 months.
  UCB4594 concentrations will be measured in serum.
Clearance of UCB4594 (monotherapy modules; Modules A and B). | From Day 1 (date of first dose of UCB4594) up to 13 months.
  UCB4594 concentrations will be measured in serum.
Frequency of AEs considered at least possibly related to UCB4594 (up to end of AE reporting period). | AEs are collected from the date of informed consent until 6 months after the last dose of UCB4594.
  The frequency of AEs will be assessed for UCB4594 (all modules) and/or other anti-cancer treatments (Module C), and the number of Grade 3, 4 and 5 AEs at least possibly related to UCB4594 (all modules) and/or other anti-cancer treatments (Module C) determined. AEs, including relatedness, seriousness and severity according to NCI CTCAE Version 5.0, will be assessed by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Thistlethwaite, Prof, Principal Investigator — The Christie NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial and the final clinical study protocol will be submitted to a public registry and will be available immediately following publication, with no end date. Individual deidentified participant data that underlie the results reported will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor. All requests made within 5 years from the end of trial will be considered; requests made subsequently will be considered where possible. Requests should be submitted to drugdev@cancer.org.uk.
Supporting Information: Study Protocol
Time Frame: Data from this trial and the final clinical study protocol will be submitted to a public registry and will be available immediately following publication, with no end date. Requests for individual deidentified participant data made within 5 years from the end of trial will be considered; requests made subsequently will be considered where possible.
Access Criteria: Individual deidentified participant data that underlie the results reported will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.

REFERENCES:
- See also: Trial registration on ISRCTN — https://www.isrctn.com/ISRCTN26628699